CLINICAL TRIAL: NCT00186485
Title: Safety and Efficacy of Open Study of Repetitive Transcranial Magnetic Stimulation (rTMS) for Treatment Resistant Bipolar Depression
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Treatment Resistant Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Hugh Brent Solvason, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stanford 79133
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-08

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Right Sided Low Frequency Unilateral TMS (Experimental): 1Hz unilateral TMS delivered to the right DLPFC using the MagStim device
  Interventions: Device: MagStim

INTERVENTIONS:
Device: MagStim — The MagStim delivers low frequency 1Hz stimulation to the right frontal area of the brain

SUMMARY:
We hope to learn whether this stimulation of neurons in the front part of the brain may relieve depression.

DETAILED DESCRIPTION:
The primary objective of this study is to examine the safety and efficacy of rTMS in the management of treatment-resistant bipolar depression.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* DSM IV Bipolar I or II Disorder with current major depressive episode
* Prior failure to respond to or tolerate at least 2 adequate pharmacotherapy trials
* Ham-D score greater than or equal to 18

Note: site enrolls only one patient per month Exclusion Criteria:Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption); b. Individuals diagnosed by the investigator with the following conditions (current unless other-wise stated): Depression secondary to a general medical condition, or substance-induced; Seasonal pattern of depression as defined by DSM-IV, History of substance abuse or dependence within the past year (except nicotine and caffeine); Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features in this or previous episodes; Obsessive compulsive disorder (lifetime); or Post-traumatic stress disorder (current or within the past year). c. An Axis II Personality Disorder, which in the judgment of the investigator may hinder the patient in completing the procedures required by the study protocol. d. Individuals with a clinically defined neurological disorder or insult including, but not limited to: Any condition likely to be associated with increased intracranial pressure; Space occupying brain lesion; Any history of seizure EXCEPT those therapeutically induced by ECT; History of cerebrovascular accident; Transient ischemic attack within two years; Cerebral aneurysm; Dementia; Mini Mental Status Exam (MMS) score of <24; Parkinson#s disease; Huntington#s chorea; or Multiple sclerosis.

e. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head trauma with loss of consciousness for >5 minutes; f. A true positive response to any question on the Transcranial Magnetic Stimulation Adult Safety Screen questionnaire (see Attachment H) g. Lifetime treatment with more than 12 antidepressant medication trials, at any dose or duration, either monotherapy or combination therapy from the list summarized in Attachment I. h. ECT treatment within 3 months prior to the screening visit; i. Failure to respond to ECT treatment (i.e., consistent with ATHF level 2 or higher) in this or any previous j. History of treatment with rTMS therapy for any disorder; k. History of treatment with Vagus Nerve Stimulation; l. Use of any investigational drug within 4 weeks of the randomization visit; m. Use of fluoxetine within 6 weeks of the randomization visit; n. Use of an MAOI within 2 weeks of the randomization visit; o. Use of any medication(s) listed on the Excluded Medication List (Attachment J) within 1 week of the randomization visit; p. Significant acute suicide risk, defined as follows: Suicide attempt within the previous 6 months that required medical treatment; or >2 suicide attempts in the past 12 months; or Has a clear-cut plan for suicide and states that he/she cannot guarantee that he/she will call his/her regular psychiatrist or the Investigator if the impulse to implement the plan becomes substantial during the study; or in the investigator#s opinion, is likely to attempt suicide within the next 6 months. q. Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease; r. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;s. Known or suspected pregnancy; t. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial; u. Positive urine drug screen. (A positive urine drug screen at screening may be repeated once prior to randomization); v. Clinically significant laboratory abnormality, in the opinion of the investigator; w. Women who are breast-feeding; x. Women of child-bearing potential not using a medically accepted form of contraception when engaging in sexual intercourse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-05; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Brent Solvason, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Right Sided Low Frequency Unilateral TMS
Started | 28
Completed | 25
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Right Sided Low Frequency Unilateral TMS: Open treatment with 1Hz unilateral TMS delivered to the right DLPFC using the MagStim device
  MagStim: The MagStim delivers low frequency 1Hz stimulation to the right frontal area of the brain
Arm/Group | Right Sided Low Frequency Unilateral TMS
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 28
Number of Subjects with Bipolar Subtype Diagnosis at Baseline [Count of Participants; unit: Participants] — The number of patients with a diagnosis of Bipolar Type I, Type II. and Not Otherwise Specified
  Participants
    Bipolar Type I | 16
    Bipolar Type II | 11
    Bipolar NOS | 1
Concurrent Medications [Number; unit: number of medications] — Medications currently taken by the patient was provided by the patient. Population: Based on a list of self-reported failed prior medication treatment trials.
  number of medications
    number analyzed (Participants) | 25
    (all) | 4
Prior Failed Medication Trials [Mean (Standard Deviation); unit: Number of medications] | 14.6 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS) -17 Item; Baseline to End of Week 4
Description: The HDRS - 17 is a scale that measures the severity of depression based on the patients response to 17 questions on the presence and severity of the symptoms found in depression. The severity of a symptom is scored from 0 (not present) to 4 (most severe); total scores range from 0 (no depressive symptoms), to 68 (very severe depression). A decrease in the HDRS score reflects a reduction in depression severity.The scores are Baseline and End of Week 4
Time Frame: 4 weeks
Population: Subjects received 4 weeks of right sided dorsolateral prefrontal cortex 1Hz TMS, last observation carried forward
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Right Sided Low Frequency Unilateral TMS
Number analyzed (Participants) | 28
units on a scale
  Baseline HDRS | 23.7 (5.9)
  End of Week 4 | 13.3 (6.0)
Statistical Analysis 1: Comparison: Right Sided Low Frequency Unilateral TMS; ANOVA with partial eta accounts for multiple repeated measures over the course of treatment; Test type: Superiority or Other; p < 0.001, ANOVA — Repeated Measures ANOVAs over the course of the TMS treatments, by severity of depression on the HAM-D rating scale: total scores (F (4,96) = 19.88, p < .001) over the 4 week treatment period; Repeated Measures Anova

2. Secondary Outcome: Beck Depression Inventory Score; Baseline to End of Week 4
Description: The Beck Depression Inventory Scale (BDI) measures the severity of depression based on the patients response to 21 questions on the presence and severity of the symptoms found in depression. The severity of a symptom is scored from 0 (not present) to 3 (most severe); total scores range from 0 (no depressive symptoms), to 63 (very severe depression). A decrease in the score reflects a reduction of the severity of depression.The scores are from Baseline and End of Week 4
Time Frame: 4 weeks
Population: Subjects received 4 weeks of right sided dorsolateral prefrontal cortex 1Hz TMS, last observation carried forward
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Right Sided Low Frequency Unilateral TMS
Number analyzed (Participants) | 28
units on a scale
  Baseline | 30.6 (7.0)
  End of week 4 | 19.4 (10.2)
Statistical Analysis 1: Comparison: Right Sided Low Frequency Unilateral TMS; Repeated measures ANOVA with partial eta; accounts for multiple repeated measures over the course of treatment; Test type: Superiority or Other; p < 0.01, ANOVA — Repeated Measures ANOVAs over the course of the TMS treatments, by severity of depression on the BDI total scores (F (4,96) = 19.35, p < .001) over the 4 week treatment period.,

3. Secondary Outcome: Clinical Global Impression - Severity; Baseline to End of Week 4
Description: The Clinical Global Impression of Severity (CGI-S) is a measure of depression severity and disability based on the clinicians overall impression of the severity of depression based on the patients response to open ended questions and self report of the presence and severity of the symptoms and level of disability found in depression. The CGI-S assesses the severity of illness (depression) and is scored from 1 (well, not at all ill) to 7 (among the most severely ill patients); a decrease in the CGI-S score reflects a reduction of the symptoms and disability due to depression. The scores are from Baseline and End of Week 4
Time Frame: 4 weeks
Population: Subjects received 4 weeks of right sided dorsolateral prefrontal cortex 1Hz TMS, last observation carried forward
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Right Sided Low Frequency Unilateral TMS
Number analyzed (Participants) | 25
units on a scale
  CGI-S baseline | 4.9 (0.68)
  CGI-S end of week 4 | 4.2 (0.83)
Statistical Analysis 1: Comparison: Right Sided Low Frequency Unilateral TMS; Repeated Measures ANOVA with partial eta; p value was adjusted for multiple comparisons over the course of treatment; Test type: Superiority or Other; p < 0.01, ANOVA — Repeated Measures ANOVAs over the course of the TMS treatments, by severity of depression on the CGI scores (F (4,88) = 5.31, p < .01) over the 4 week treatment period

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Right Sided Low Frequency Unilateral TMS
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 6/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Right Sided Low Frequency Unilateral TMS (N=28)
mild headache (Musculoskeletal and connective tissue disorders) | 6 (6) — transient headache in the area of TMS stimulation. Resolved shortly after treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes